CLINICAL TRIAL: NCT06494397
Title: Crossover Bioequivalence Study of 12 mg VHX-896 and Iloperidone Tablets Under Steady-State Conditions
Brief Title: Pharmacokinetic Study of VHX-896 and Iloperidone Tablets Under Steady-State Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VP-VHX-896-1103
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: Iloperidone; VHX-896
MeSH Terms: conditions — Schizophrenia | interventions — iloperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: VHX-896 then iloperidone (Experimental)
  Interventions: Drug: VHX-896 and iloperidone
- Sequence B: Iloperidone then VHX-896 (Experimental)
  Interventions: Drug: Iloperidone and VHX-896

INTERVENTIONS:
Drug: VHX-896 and iloperidone — oral tablet
  Arms: Sequence A: VHX-896 then iloperidone
Drug: Iloperidone and VHX-896 — oral tablet
  Arms: Sequence B: Iloperidone then VHX-896

SUMMARY:
Study to compare the pharmacokinetics and pharmacodynamics of VHX-896 and iloperidone and evaluate the safety and tolerability of VHX-896 and iloperidone in patients with schizophrenia or bipolar I disorder under steady state conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 to 65 years of age (inclusive)
* Diagnosed with either schizophrenia or bipolar I disorder, manic or mixed type, according to the Diagnostic and Statistical Manual of Mental Disorder, Fifth Edition, Text Revision (DSM-5-TR)
* Patients must be symptomatically stable and on a stable treatment with an oral atypical antipsychotic at an adequate dose (3 months prior to enrollment) and not suffer from acute increase of their psychosis or be hospitalized within the past 2 months

Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Cytochrome P450 2D6 (CYP2D6) poor metabolizers and use of prescription medication or OTC medication that strongly inhibits CYP2D6 or CYP3A4 or induces CYP3A4 within 5 half-lives of baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Bioequivalence between VHX-896 tablets relative to iloperidone tablets | 12 hours
  As measured by plasma concentrations

SECONDARY OUTCOMES:
Assessment of safety and tolerability of VHX-896 and iloperidone | 24 days
  As measured by spontaneous reporting of adverse events (AEs).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Vanda Investigational Site, Los Alamitos, California
  - Vanda Investigational Site, Gaithersburg, Maryland
  - Vanda Investigational Site, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No